CLINICAL TRIAL: NCT01828762
Title: Clinical Study of the Safety of Autologous Immune Cell Therapy in Primary Hepatocellular Carcinoma Patients Following Resection and TACE Therapy
Brief Title: Autologous Immune Cell Therapy in Primary Hepatocellular Carcinoma Patients Following Resection and TACE Therapy
Acronym: DC-TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: No.85 Hospital, Changning, Shanghai, China (Other); China Cell Technology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040420100005
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-04

CONDITIONS: Primary Hepatocellular Carcinoma
Keywords: DC; Immunotherapy; TC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC-TC+GM-CSF (Experimental)
  Interventions: Biological: DC-TC+GM-CSF

INTERVENTIONS:
Biological: DC-TC+GM-CSF

SUMMARY:
Although liver resection, liver transplantation, a-interferon, Transarterial Chemo Embolization (TACE), percutaneous ethanol injection (PEI), Percutaneous microwave coagulation therapy (PMCT), Radiofrequency ablation (RFA) provide options to treat patients with HCC, the high recurrence rate of mid-late stage liver cancer still exists. The safety of autologous Immune Cell Therapy in Primary Hepatocellular Carcinoma (HCC) Patients Following Resection and TACE Therapy will be evaluated.

DETAILED DESCRIPTION:
The study is a single center,open label trial. To obtain safety information on toxicities and adverse events attributable to the subcutaneous injections of autologous dendritic cells incubated with irradiated autologous tumor stem cells and suspended in GM-CSF in patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent signed by patient or legal guardian, obtained prior to study enrollment.
2. BCLC Classification A-B
3. Patients who are good surgical candidates for HCC resection
4. ECOG Performance Score, 0-1
5. Child-Pugh Rating, A
6. Expected survival greater than 6 months

Exclusion Criteria:

1. History of anaphylactic reaction to GM-CSF
2. Congestive heart failure, unstable angina or other underlying cardiac disease; history of thrombosis currently requiring anticoagulation
3. Mental or psychological illness preventing cooperation with treatment, efficacy evaluations, or unable to understand the informed consent process
4. Primary cancers of any kind or location, other than hepatocellular carcinoma
5. Excluding hepatitis, any active or unresolved infection including HIV, EBV, CMV, RPR, TB, etc.
6. Autoimmune disease requiring therapy; immunodeficiency, or any disease process requiring immunosuppressive therapy.
7. Prior clinical trial requiring patient to receive an investigational drug within two weeks of enrollment.
8. Pregnant or lactating women.
9. Patients with the intention to receive transplantation
10. Significant comorbidity or other active medical condition that could be eminently life threatening in the opinion of the investigator, including no active blood clotting or bleeding diathesis.
11. Evidence of metastatic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Vital signs，physical examinations and adverse events | one year
  The number of adverse events along with the results of vital signs measurements, physical examinations, and clinical laboratory tests will be used to determine the safety profile of DC-TC.

CONTACTS AND LOCATIONS:
Overall Officials: Chengwei Chen, Principal Investigator — No.85 Hospital, Changning, Shanghai, China
Locations (1):
- 9585 Humin Road,Xuhui district, Shanghai, Shanghai Municipality, China